CLINICAL TRIAL: NCT00403338
Title: Prospective Evaluation of the Impact of Stent Deployment Techniques on Clinical Outcomes of Patient Treated With the CYPHER® Stent, The e-CYPHER(SM)S.T.L.L.R., Registry [Study of Deployment Technique on Clinical Results]
Brief Title: The Impact of Stent Deployment Techniques on Clinical Outcomes of Patient Treated With the CYPHER® Stent (S.T.L.L.R.)
Status: Completed | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Other Study IDs: P03-6323
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Coronary Stenosis
Keywords: myocardial ischemia; coronary disease; heart disease; Coronary Stenosis [MeSH heading: C14.280.647.250.285]
MeSH Terms: conditions — Coronary Stenosis; Myocardial Ischemia; Coronary Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CYPHER® Bx Velocity™ stent (sirolimus-eluting)

SUMMARY:
1500 eligible patients will be treated with the commercially available CYPHER® sirolimus-eluting Bx Velocity™ stent. Patients will be followed to twelve months post-procedure, watching for patients that require a repeat procedure on the same diseased area of the coronary artery.

DETAILED DESCRIPTION:
Geographical miss has been associated with treatment failures after intracoronary radiation therapy. This phenomenon, which is secondary to vascular injury outside the treated segment, was strongly correlated with the development of restenosis at the edges of the treated coronary segment. The European and Canadian SIRIUS trials (E and C-SIRIUS) randomized 350 patients with similar baseline characteristics of the US SIRIUS study. Operators used shorter post-dilatation balloons and direct stented 27% of the patients, achieving a 4.0% TLR rate and a 5.1% in-lesion binary restenosis. These somewhat superior results support the concept that refinement in deployment techniques may further improve clinical outcomes of drug-eluting stents.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of de novo stenosis in major coronary artery
* Can be treated with stents
* Candidate for bypass

Exclusion criteria:

* Recent, severe MI
* Prior brachytherapy
* Impaired left ventricle function
* Heart transplant recipient
* Impaired renal function
* Disease in vein grafts from previous bypass
* Similar treatment within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing an intervention and receiving a CYPHER stent.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2004-12; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Orlick, Study Director — Cordis Corporation, a Johnson & Johnson Co.

REFERENCES:
- [Result] Costa MA, Angiolillo DJ, Tannenbaum M, Driesman M, Chu A, Patterson J, Kuehl W, Battaglia J, Dabbons S, Shamoon F, Flieshman B, Niederman A, Bass TA; STLLR Investigators. Impact of stent deployment procedural factors on long-term effectiveness and safety of sirolimus-eluting stents (final results of the multicenter prospective STLLR trial). Am J Cardiol. 2008 Jun 15;101(12):1704-11. doi: 10.1016/j.amjcard.2008.02.053. Epub 2008 Apr 9. PMID 18549844
- [Result] Suzuki N, Angiolillo DJ, Tannenbaum MA, Driesman MH, Smith C, Bikkina M, Meckel CR, Morales CE, Xenopoulos NP, Coletta JE, Bezerra HG, Bass TA, Costa MA. Strategies for drug-eluting stent treatment of bifurcation coronary artery disease in the United States: insights from the e-Cypher S.T.L.L.R.trial. Catheter Cardiovasc Interv. 2009 Jun 1;73(7):890-7. doi: 10.1002/ccd.21796. PMID 19455662